CLINICAL TRIAL: NCT03745248
Title: Effects of Aerobic Exercise on Degenerative Cerebellar Disease
Brief Title: Aerobic Exercise, Balance Training, and Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Joel Stein, MD, Clinical investigator, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAR5381
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Ataxia; Spino Cerebellar Degeneration; Spinocerebellar Ataxias
Keywords: Degenerative cerebellar disease; Ataxia; Aerobic Exercise
MeSH Terms: conditions — Ataxia; Spinocerebellar Degenerations; Spinocerebellar Ataxias

STUDY DESIGN:
Intervention Model Description: Single blind randomized control trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will know that the participant has received balance or aerobic training, but will not be aware of which group the participant belonged
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Training (Experimental): Participants will be given a stationary exercise bike for home use. They will be instructed to use the exercise bike five times a week for thirty-minute sessions. The exercise intensity prescription will be based on the subject's VO2max determined on pre-test day. The exercise program will start at 60% of intensity per session, and then will be increased by steps of 5% intensity every 2 sessions until participants reach 30 minutes of training at 80% intensity. Participants will be contacted weekly by e-mail or phone to answer any questions about the exercise protocol and will be instructed to log each training session. Subjects will record duration of exercise, perceived exertion, average heart rate, maximum heart rate, and distance.
  Interventions: Behavioral: Aerobic training
- Balance Training (Active Comparator): A physical therapist will tailor a home balance training program for each participant based on pre-training capabilities. Subjects will be asked to perform exercises five times a week for thirty-minute sessions. Both dynamic and static exercises will be performed in sitting and standing positions. Exercises will start with stabilizing in a challenging static position and progress to dynamic arm and leg movements in the same or modified position. Participants will be contacted weekly by e-mail or phone to answer any questions about the exercise protocol and will be required to log their exercise effort in terms of frequency and level of balance challenge. Individuals will be instructed to perform more difficult exercises if balance challenge scores are low.
  Interventions: Behavioral: Balance Training

INTERVENTIONS:
Behavioral: Aerobic training — Aerobic training on stationary bicycle for 30 minutes a day, 5 days a week for 1 month
  Arms: Aerobic Training
Behavioral: Balance Training — Standard of care
  Arms: Balance Training

SUMMARY:
The first aim is to show aerobic training improves degenerative cerebellar patients functionally

The second aim is to compare the effects of balance and aerobic training on degenerative cerebellar disease.

DETAILED DESCRIPTION:
Individuals with degenerative cerebellar disease (DCD) exhibit gradual loss of coordination resulting in impaired balance, gait deviations, and severe, progressive disability. With no available disease-modifying medications, balance training is the primary treatment option to improve motor skills and functional performance.

Aerobic training, on the other hand, may modify DCD progression as evident from animal data. Compared to sedentary controls, aerobically trained DCD rats have enhanced lifespan, motor function, and cerebellar Purkinje cell survival. Numerous animal studies also document that aerobic training has a direct, favorable effect on the brain that includes production of neurotrophic hormones, enhancement of neuroplasticity mechanisms, and protection from neurotoxins.

The effects of aerobic training in humans with DCD are relatively unknown, despite these encouraging animal data. A single study to date has evaluated the benefits of aerobic exercise on DCD in humans, and this was a secondary outcome of the study. Although participants performed limited aerobic training during the study, modest functional benefits were still detected.

The main objective of this project will be to compare the benefits of aerobic versus balance training in DCD. The investigators hypothesize that both aerobic and balance training will improve function in DCD subjects, but that the mechanisms in which these improvements occur differ.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spinocerebellar ataxia
* Cerebellar atrophy on MRI
* Prevalence of ataxia on clinical exam
* Ability to safely ride a stationary exercise bike

Exclusion Criteria:

* Other neurologic conditions
* Heart disease
* Cognitive impairment
* Medical instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-06-09 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Change in SARA score | 1 month
  Ataxia severity will be measured using the Scale for the Assessment and Rating of Ataxia (SARA).SARA evaluates the degree of ataxia by measuring gait, stance, sitting balance, speech, finger-chase test, nose-finger test, fast alternating movements, and heel-shin test.

SECONDARY OUTCOMES:
Change in gait speed | 1 month
  For the walking assessment, participants will walk as fast as possible on a 10-meter runway six times, and the investigators will average the times of trials 3-6 to determine gait speed expressed in meters/second.
Change in static balance | 1 month
  Static standing balance will be assessed by measuring postural sway during two, one-minute trials. Participants will stand with arms crossed over their chest and feet shoulder-width apart under two conditions: eyes open and eyes closed. Data will be collected using Bertec's dual split-belt treadmill (Bertec, Columbus, OH) embedded with force plates. Balance deficits will be calculated as the magnitude of postural sway (sway amplitude) using custom Nexus and Bodybuilder software (Vicon, Denver, CO).

CONTACTS AND LOCATIONS:
Overall Officials: Joel Stein, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University/New York Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barbuto S, Martelli D, Isirame O, Lee N, Bishop L, Kuo SH, Agrawal S, Lee S, O'Dell M, Stein J. Phase I Single-Blinded Randomized Controlled Trial Comparing Balance and Aerobic Training in Degenerative Cerebellar Disease. PM R. 2021 Apr;13(4):364-371. doi: 10.1002/pmrj.12401. Epub 2020 May 29. PMID 32383352